CLINICAL TRIAL: NCT01344889
Title: Global Observational Cohort Study on the Prediction of Unwanted Adverse Effects in Individuals Infected With Chronic Hepatitis C Receiving a Long Acting Interferon Plus Ribavirin
Brief Title: An Observational Study on The Prediction of Adverse Events in Patients With Chronic Hepatitis C Receiving a Long-Acting Interferon Plus Ribavirin (GUARD-C)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MV22255
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess factors leading to dose reductions/treatment discontinuations and the effect on sustained virological response in patients with chronic hepatitis C receiving a long-acting interferon (e.g. Pegasys/peginterferon alfa-2a) and ribavirin. Data will be collected from each patient for the duration of their treatment and for up to 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (according to local legislation)
* Chronic hepatitis C
* Treatment with long-acting interferon plus ribavirin
* Quantifiable HCV RNA before initiation of treatment
* No contra-indications to long-acting interferon and ribavirin therapy as detailed in the label

Exclusion Criteria:

* End stage renal disease
* Major organ transplantation
* Concomitant therapy with telbivudine
* Pregnant or breast-feeding females
* Male partners of pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C receiving a long-acting interferon plus ribavirin
Sampling Method: Probability Sample
Enrollment: 4459 (Actual)
Dates: Start 2009-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Correlation between baseline patient characteristics and safety related dose reductions/treatment discontinuations of the long-acting interferon or ribavirin | 4 years
Correlation between safety related dose reductions/treatment discontinuations and sustained virological response (SVR: defined as HCV RNA <50 IU/mL at 24 weeks after completion of treatment) | 4 years

SECONDARY OUTCOMES:
Correlation of on-treatment factors and dose reduction/treatment discontinuation | 4 years
Correlation between degree of dose reductions/treatment interruptions (percentage of actual exposure/treatment administrations in relation to target exposure) and SVR | 4 years
Comparison of on-treatment virological response (rapid virological response, early virological response) in treatment-naïve and treatment experienced patients | 4 years
Safety: Incidence of adverse events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (192):
- Albania (2):
  - Elbasan
  - Tirana
- Algiers, Algeria
- Bahrain (2):
  - Bahrain
  - Manama
- Belgium (20):
  - Antwerp
  - Bruges
  - Brussels
  - Charleroi
  - Edegem
  - Genk
  - Gerrardsbergen
  - Ghent
  - Haine-Saint-Paul
  - Hasselt
  - Kortrijk
  - Leuven
  - Liège
  - Mont-godinne
  - Namur
  - Ostend
  - Roeselare
  - Seraing
  - Sijsele
  - Verviers
- Bosnia and Herzegovina (6):
  - Banja Luka
  - Bihać
  - Mostar
  - Sarajevo
  - Tuzla
  - Zenica
- Brazil (12):
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Uberaba, Minas Gerais
  - Nova Iguaçu, Rio de Janeiro
  - Rio de Janeiro, Rio de Janeiro
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Santo André, São Paulo
  - Santos, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Egypt (3):
  - Alexandria
  - Cairo
  - Tanta
- Greece (7):
  - Alexandroupoli
  - Athens
  - Ioannina
  - Pátrai
  - Piraeus
  - Rhodes
  - Thessaloniki
- Hungary (20):
  - Ajka
  - Balassagyarmat
  - Békéscsaba
  - Budapest
  - Debrecen
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Miskolc
  - Mosonmagyaróvár
  - Nyíregyháza
  - Pécs
  - Sopron
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Zalaegerszeg
- India (8):
  - Pune, Maharashtra
  - Hyderabad
  - Kochi
  - Lucknow
  - Ludhiana
  - Mizoram
  - Mumbai
  - Noida
- Tehran, Iran
- Italy (46):
  - Pescara, Abruzzo
  - Brindisi, Apulia
  - Foggia, Apulia
  - Galatina, Apulia
  - San Giovanni Rotondo, Apulia
  - Catanzaro, Calabria
  - Reggio Calabria, Calabria
  - Avellino, Campania
  - Benevento, Campania
  - Gragnano, Campania
  - Napoli, Campania
  - Salerno, Campania
  - Bologna, Emilia-Romagna
  - Carpi, Emilia-Romagna
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Ravenna, Emilia-Romagna
  - Udine, Friuli Venezia Giulia
  - Frosinone, Lazio
  - Gaeta, Lazio
  - Rome, Lazio
  - Genoa, Liguria
  - Brescia, Lombardy
  - Busto Arsizio, Lombardy
  - Como, Lombardy
  - Milan, Lombardy
  - Treviglio, Lombardy
  - Campobasso, Molise
  - Asti, Piedmont
  - Biella, Piedmont
  - Novara, Piedmont
  - Omegna (VB), Piedmont
  - Orbassano, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Comiso, Sicily
  - Messina, Sicily
  - Palermo, Sicily
  - Torrette Di Ancona, The Marches
  - Florence, Tuscany
  - Pisa, Tuscany
  - Perugia, Umbria
  - Padua, Veneto
  - Rovigo, Veneto
- Kuwait (2):
  - Hawali
  - Safat
- Lebanon (4):
  - Baabda
  - Beirut
  - Saida
  - Tripoli
- Morocco (2):
  - Casablanca
  - Rabat
- Skopje, North Macedonia
- Pakistan (5):
  - Faisalabad
  - Hyderābād
  - Karachi
  - Lahore
  - Rawalpindi
- Poland (16):
  - Bialystok
  - Bydgoszcz
  - Bytom
  - Chorzów
  - Cieszyn
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Puławy
  - Racibórz
  - Tychy
  - Warsaw
  - Wałbrzych
  - Wroclaw
  - Łańcut
- Portugal (10):
  - Almada
  - Amadora
  - Aveiro
  - Beja
  - Coimbra
  - Faro
  - Lisbon
  - Porto
  - Santarém
  - Vila Real
- Doha, Qatar
- Romania (7):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Craiova
  - Iași
  - Timișoara
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Sad
- Slovakia (6):
  - Banská Bystrica
  - Bratislava
  - Košice
  - Martin
  - Prešov
  - Trenčín
- South Korea (4):
  - Buchun
  - Busan
  - Seoul
  - Suwon
- United Arab Emirates (2):
  - Abu Dhabi
  - Dubai

REFERENCES:
- [Derived] Foster GR, Coppola C, Derbala M, Ferenci P, Orlandini A, Reddy KR, Tallarico L, Shiffman ML, Ahlers S, Bakalos G, Hassanein T; GUARD-C Study Group. Impact of Safety-Related Dose Reductions or Discontinuations on Sustained Virologic Response in HCV-Infected Patients: Results from the GUARD-C Cohort. PLoS One. 2016 Mar 28;11(3):e0151703. doi: 10.1371/journal.pone.0151703. eCollection 2016. PMID 27018988